CLINICAL TRIAL: NCT03977090
Title: Phase Ib Clinical Trial of Geptanolimab Combined With Fruquintinib in the Treatment of Metastatic Colorectal Cancer
Brief Title: Geptanolimab(GB226) Combined With Fruquintinib in the Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-012-1
Record Dates: First submitted 2019-05-24; First posted 2019-06-06 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB226+Fruquintinib (Experimental): Geptanolimab combined with Fruquintinib
  Interventions: Drug: Geptanolimab Injection; Drug: Fruquintinib

INTERVENTIONS:
Drug: Geptanolimab Injection — GB226 3mg/kg, q2w, iv.
  Other Names: Recombinant humanized anti-PD-1 monoclonal antibody injection; Geptanolimab
Drug: Fruquintinib — Fruquintinib 3 or 4 or 5mg,qd,po. 3 weeks-on, 1 week-off
  Other Names: HMPL-013

SUMMARY:
This study is a multicenter, dose-escalating phase Ib clinical study to evaluate the safety and tolerability of GB226 in combination with fruquintinib in the treatment of mCRC, evaluate the pharmacokinetic characteristics of GB226 in combined therapy, evaluate immunogenicity of GB226, and explore the antitumor activity of GB226 in combination with fruquintinib in the treatment of mCRC.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria can be enrolled in this study:

1. Aged 18 to 75 years, males or females;
2. Understand the study procedures and contents, and voluntarily sign the written informed consent form;
3. Patients with histologically/pathologically confirmed colorectal cancer;
4. Patients with metastatic colorectal cancer, who failed to respond to the previous first-line treatment or above. Treatment failure refers to disease progression or intolerable toxicity after ≥1 cycle of treatment, or relapse during adjuvant or neoadjuvant chemotherapies period or within 6 months after the end of treatment;
5. ECOG score of 0-1;
6. Life expectancy≥3 months;
7. There is at least one measurable and evaluable tumor lesion (in accordance with RECIST1.1 criteria);
8. Systemic chemotherapy, targeted therapies or other anti-tumor biotherapy (tumor vaccine, cytokine or growth factor aimed at controlling tumor) are completed at least 4 weeks before the first dose of investigational product (the oral fluorouracil is discontinued at least 2 weeks ago); systemic or local palliative radiotherapy is completed at least 4 weeks ago; no anti-angiogenic small molecular target drugs are previously received;
9. Systemic corticosteroids (prednisone > 10mg/day or equivalent dose) is discontinued at least 2 weeks before the use of the first investigational product;
10. The major surgery requiring general anesthesia must be completed at least 8 weeks before the use of the first investigational product; surgery requiring local anesthesia/epidural anesthesia must be completed at least 4 weeks before the use of the first investigational product;
11. Routine blood tests require hemoglobin (HGB) ≥90g/L (no transfusion is allowed within 14 days before routine blood tests at baseline), neutrophil count (ANC)≥1.5×109/L (received no supportive treatment with recombinant human granulocyte colony stimulating factor within 14 days before routine blood tests at baseline), platelet ≥100×109/L (received no supportive treatment such as recombinant human thrombopoietin (TPO) or transfusion within 14 days before routine blood tests at baseline);
12. Serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 60 mL/min (calculated based on Cockcroft-Gault formula), and urinary protein ˂ 2+ or ˂1.0g/L; For patients with baseline urinary protein ≥ 2+ or ≥ 1.0g/L, quantitative test of 24h urinary protein will be performed and will be enrolled only when the result ≤ 1.0g/L is obtained.
13. Total bilirubin ≤1.5×ULN (unless it is confirmed to have Gilbert's Syndrome), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (AST and/or ALT≤5×ULN is allowed for patients with hepatic metastasis);
14. Thyroid function variables: thyroid-stimulating hormone (TSH) and free thyroxine (FT3/FT4) are within the normal range; if TSH is not within the normal range, but FT3/FT4 is within the normal range, the subjects can be enrolled.
15. The adverse reactions caused by the previous treatment should recover to grade 1 and below before enrollment (except alopecia and ≤ grade 2 neurological toxicity caused by chemotherapy drugs);
16. Female subjects who are confirmed not pregnant within 7 days before administration; males or females should agree to adopt medically confirmed effective contraceptive measures during the entire study period and within 6 months after the end of this study.
17. Patients can receive follow-up visits as scheduled, well communicate with the investigators and complete the study as required by the study.

Exclusion Criteria:

Any patient fulfilling any of the following exclusion criteria is excluded from this study:

1. Active central nervous system (CNS) metastasis, including symptomatic brain metastasis or meningeal metastasis or spinal cord compression etc.; subjects with asymptomatic brain metastasis (no progression within at least 4 weeks after radiotherapy and/or no neurological symptom or sign after surgical resection, treatment with glucocorticoids, antiepileptic drugs, anticonvulsants or mannitol is not necessary) can be enrolled;
2. Patients who previously had other malignant tumors (excluding cured cervical carcinoma in situ and skin basal cell carcinoma) are not allowed to participate in the study unless he/she completely relieved at least 2 years before enrollment and requires no other treatment now or during the study period.
3. Medical history of active, known autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory gastrointestinal disorders, Hashimoto's thyroiditis etc. The following should be excluded: type I diabetes mellitus, hypothyroidism which can be controlled by hormone replacement therapies only, skin diseases requiring no systemic treatment (e.g., vitiligo, psoriasis) and controlled celiac disease;
4. Patients who are previously treated with anti PD-1 antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4 antibody (or any other antibodies acting on T cell co-stimulation or checkpoint pathway);
5. Uncontrolled hypertension ( systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) or pulmonary arterial hypertension or unstable angina pectoris; previous presence of myocardial infarction or received coronary artery bypass grafting or coronary stent implantation within 6 months before administration; medical history of chronic heart failure NYHA (New York Heart Association) class 3 and 4; clinically significant valvular heart diseases; subjects with serious arrhythmia requiring treatment, including QTc interval ≥450ms for males and ≥470ms for females (calculated based on Fridericia formula); cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 months before administration;
6. Patients who have medical history of arterial thrombosis or deep vein thrombosis within 6 months before the first dose of investigational product, or patients who have evidence or medical history of bleeding tendency within 2 months before the first dose of investigational product, regardless of severity; activated partial thromboplastin time (APTT) or prothrombin time (PT) >1.5×ULN;
7. The skin wounds, surgery site, trauma site, serious mucosal ulcer or facture are not completely healed.
8. The imaging tests showing the evidence of tumor invasion to large vessels, including tumors which are completely close to, surround or invade to internal cavity of large vessels (e.g., pulmonary artery or superior vena cava);
9. Patients with dysphagia or known drug malabsorption;
10. Gastrointestinal disorder which may significantly affect absorption of oral drugs or other conditions which may affect gastrointestinal hemorrhage or perforation (e.g., duodenal ulcer, bowel obstruction, acute Crohn's disease, ulcerative colitis, resection of large area of stomach and small intestine etc.) at the discretion of the investigators; Patients who have chronic Crohn's disease and ulcerative colitis (excluding patients with resection of entire colon and rectum), even in non-active stage, should be excluded. Patients with hereditary nonpolyposis colorectal cancer or familial adenomatous polyposis syndrome; Previous medical history of intestinal perforation, intestinal fistula, which is not cured after surgical treatment;
11. Subjects with current or previous interstitial lung pneumonia;
12. Uncontrolled pleural, peritoneal and pericardial effusion requiring repeated drainage or showing significant symptoms;
13. Patients with active infection requiring systemic treatment; active pulmonary tuberculosis (TB) infection;
14. Positive human immunodeficiency virus antibody (HIV-Ab); active syphilis; positive hepatitis C antibody (HCV-Ab) and HCV-RNA> the upper limit of normal of the test units; positive hepatitis B surface antigen (HBsAg) and HBV-DNA copies > the upper limit of normal of the test units;
15. Patients with complications requiring treatment with immunosuppressive drugs or systemic or local corticosteroids at the immunosuppressive doses (prednisone > 10mg/day or equivalent dose of similar agents);
16. It is expected that live vaccines or attenuated vaccines are given 4 weeks before the use of investigational drug, during treatment period or within 5 months after the last dose;
17. Subjects who have medical history of drug addiction or drug abuse;
18. Lactating women (subjects who agree to stop breastfeeding during the study period can be enrolled);
19. Patients who received other investigationsl drugs within 30 days before the use of investigational drug or within 5 half-lives of other investigational drugs (whichever is shorter) or used investigational medical device within 30 days;
20. Subjects who are known to be allergic to investigational product or any of its excipients; subjects who are known to have medical history of allergic diseases;
21. Subjects who are considered unsuitable for participating in this study at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | up to 52 weeks
  Adverse Event
Dose Limited Toxicity,DLT | up to 52 weeks
  To evaluate the safety of GB226 as defined by dose limited toxicity in patients with metastatic colorectal cancer.
Extended period recommended dose,RDE | up to 52 weeks
  To evaluate the safety of GB226 as defined by extended period recommended dose in patients with metastatic colorectal cancer.

SECONDARY OUTCOMES:
T max | up to 52 weeks
  T max
C max | up to 52 weeks
  C max
C ss,min | up to 52 weeks
  C ss,min
R C,trough | up to 52 weeks
  R C,trough
Objective Response Rate, ORR | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by objective response rate in patients with metastatic colorectal cancer.
Disease control rate (DCR) | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by overall response rate, in patients with metastatic colorectal cancer.
Duration of response, DOR | up to 52 weeks
  To evaluate the duration of response (DOR) of GB242 in patients with metastatic colorectal cancer.
Progression-free survival, PFS | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by progression-free survival in patients with metastatic colorectal cancer.
Overall survival, OS | up to 52 weeks
  To evaluate the duration from the first administration to death because of any reason in patients with metastatic colorectal cancer.
Antidrug antibody, ADA | up to 52 weeks
  Antidrug antibody, ADA

CONTACTS AND LOCATIONS:
Overall Officials: Yuxian Bai, Principal Investigator — Affiliated tumor hospital of Harbin medical university
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No